CLINICAL TRIAL: NCT05546567
Title: NOPARK Open Label Extension Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 457567
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Safety Issues
Keywords: Parkinson's disease; Nicotinamide Riboside; Open Label
MeSH Terms: conditions — Parkinson Disease | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: Open label single group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nicotinamide Riboside (Experimental): Open Label. Nicotinamide Riboside 1200mg x1 daily
  Interventions: Dietary Supplement: Nicotinamide Riboside

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside — 1200mg x1 Nicotinamide Riboside

SUMMARY:
This protocol describes the NOPARK Open Label Extension Study. The NOPARK Open Label Extension study is an optional extension of the clinical phase II NOPARK study. Participants who have been included in the NOPARK study will upon completing their participation in the NOPARK study (i.e., after 52 weeks) be offered to receive the study drug Nicotinamide Riboside (NR) 1200 mg P.O. per day, until the NOPARK trial is completed, and the data analyzed with a conclusion of the primary outcome. Individuals enrolled into the NOPARK Open Label Extension Study will be followed with yearly visits. The goal of the NOPARK Open Label Extension Study is to monitor long term safety and study long term neuroprotective and other biological effects of NR use.

DETAILED DESCRIPTION:
The primary objective of the NOPARK open label extension study is to monitor NR use for long term safety. The secondary objective of the NOPARK open label study is to monitor long term NR use among PD patients and observe the clinical progression of PD. The NOPARK open label extension study is an open label study, where subjects enrolled in the NOPARK study (ClinicalTrials.gov: NCT03816020), upon completion of the study, will be offered the NR study drug for continuous use, until the NOPARK study is completed and the primary end-point assessed (31/12/2025). The dose of NR is 1200mg NR daily, divided into 600mg twice daily. The reason for the slightly higher dose compared to NOPARK (i.e., 200mg higher) is the fact that the active compound is now available in capsules of 300mg which cannot be divided. From a clinical and scientific perspective, given current knowledge of safety and efficacy of NR in PD, a dose of 1200 mg is both safe and of a higher potential benefit to patients. The study is multi-site, identical to NOPARK. The primary endpoint of the study, which is safety, will be analyzed using descriptive statistics. The secondary endpoint, which is if long-term NR use delays PD progression will be analyzed using the clinical MDS-UPDRS score. Exploratory objectives will assess PD progression relative to the general PD-population and whether long-term NR use affects methylation metabolism. Stratification of analyses is dependent on the duration of administered NR, sex and age. Exploratory stratification will be done based on results from biological data analysis based on data from NOPARK or blood samples collected in the NOPARK open label extension study.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form

Stated willingness to comply with all study procedures and availability for the duration of the study

Participated in the NOPARK study

Exclusion Criteria:

* Current use of vitamin B3 supplementation or NR supplementation - other than in relation to the NOPARK study

Known allergic reactions to components of the NR

Physical or psychiatric illness that makes them unavailable for follow-up and participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Safety: measurement of Adverse Events | 0-3 Years
  To assess the safety profile of long-term treatment with oral NR 1200 mg daily.

SECONDARY OUTCOMES:
Clinical Outcome: total movement disorders society unified Parkinson disease rating scale (MDS-UPDRS) score. Range 0-199 | 0-3 Years
  To assess whether the progression of PD during the NOPARK open label extension study differs among individuals who used placebo and individuals who used NR for 52 weeks in the NOPARK study.

CONTACTS AND LOCATIONS:
Overall Officials: Charalampos Tzoulis, PhD, Principal Investigator — Neur-Sysmed, Haukeland University Hospital, Norway
Locations (1):
- Haukeland University Hospital, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: Yes
All data supporting te publication will be publicly shared with the exception of any sensitive information which can lead to participant identification, as defined by Norwegian law.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At publication
Access Criteria: We will publish open access. The data will be publicly available

REFERENCES:
- [Background] Brakedal B, Dolle C, Riemer F, Ma Y, Nido GS, Skeie GO, Craven AR, Schwarzlmuller T, Brekke N, Diab J, Sverkeli L, Skjeie V, Varhaug K, Tysnes OB, Peng S, Haugarvoll K, Ziegler M, Gruner R, Eidelberg D, Tzoulis C. The NADPARK study: A randomized phase I trial of nicotinamide riboside supplementation in Parkinson's disease. Cell Metab. 2022 Mar 1;34(3):396-407.e6. doi: 10.1016/j.cmet.2022.02.001. PMID 35235774
- [Background] Dollerup OL, Christensen B, Svart M, Schmidt MS, Sulek K, Ringgaard S, Stodkilde-Jorgensen H, Moller N, Brenner C, Treebak JT, Jessen N. A randomized placebo-controlled clinical trial of nicotinamide riboside in obese men: safety, insulin-sensitivity, and lipid-mobilizing effects. Am J Clin Nutr. 2018 Aug 1;108(2):343-353. doi: 10.1093/ajcn/nqy132. PMID 29992272
- [Background] Conze DB, Crespo-Barreto J, Kruger CL. Safety assessment of nicotinamide riboside, a form of vitamin B3. Hum Exp Toxicol. 2016 Nov;35(11):1149-1160. doi: 10.1177/0960327115626254. Epub 2016 Jul 11. PMID 26791540
- [Background] Conze D, Brenner C, Kruger CL. Safety and Metabolism of Long-term Administration of NIAGEN (Nicotinamide Riboside Chloride) in a Randomized, Double-Blind, Placebo-controlled Clinical Trial of Healthy Overweight Adults. Sci Rep. 2019 Jul 5;9(1):9772. doi: 10.1038/s41598-019-46120-z. PMID 31278280
- [Background] EFSA Panel on Nutrition, Novel Foods and Food Allergens (NDA); Turck D, Bohn T, Castenmiller J, De Henauw S, Hirsch-Ernst KI, Maciuk A, Mangelsdorf I, McArdle HJ, Naska A, Pelaez C, Pentieva K, Siani A, Thies F, Tsabouri S, Vinceti M, Cubadda F, Frenzel T, Heinonen M, Prieto Maradona M, Marchelli R, Neuhauser-Berthold M, Poulsen M, Schlatter JR, van Loveren H, Albert O, de Sesmaisons Lecarre A, Knutsen HK. Extension of use of nicotinamide riboside chloride as a novel food pursuant to Regulation (EU) 2015/2283. EFSA J. 2021 Nov 12;19(11):e06843. doi: 10.2903/j.efsa.2021.6843. eCollection 2021 Nov. PMID 34804232